CLINICAL TRIAL: NCT06139172
Title: Promoting Prosocial Behavior in Syndromic Intellectual and Developmental Disabilities
Brief Title: Web Intervention for Parents of Youth With Genetic Syndromes (WINGS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Latha Soorya, Associate Professor | Department of Psychiatry & Behavioral Sciences Director | AARTS Center, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21012004
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Telomeric 22Q13 Monosomy Syndrome; Tuberous Sclerosis; Hamartoma Syndrome, Multiple; Fragile X Syndrome; Angelman Syndrome; Rett Syndrome; Chromosome 15Q, Partial Deletion; Creatine Deficiency, X-linked
MeSH Terms: conditions — Telomeric 22q13 Monosomy Syndrome; Tuberous Sclerosis; Hamartoma Syndrome, Multiple; Fragile X Syndrome; Angelman Syndrome; Rett Syndrome; Chromosome 15q, partial deletion; Creatine deficiency, X-linked

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Behavioral Training (Experimental)
  Interventions: Behavioral: Functional Behavioral Training (FBT)
- Positive Parenting Strategies-Treatment As Usual (Active Comparator)
  Interventions: Other: Positive Parenting Strategies-Treatment as Usual

INTERVENTIONS:
Behavioral: Functional Behavioral Training (FBT) — Function-based treatment (FBT) is a term for behavioral intervention approaches that use objective and systematic data collection to identify the cause of challenging behavior and teach a more prosocial replacement behavior. FBTslDD incorporates standard elements of FBT protocols with adaptations made specifically to support application to the syndromic IDD population. FBTslDD will include the following steps: (1) Syndromic IDD screening; (2) Stimulus preference assessment; (3) Indirect and descriptive assessments; (4) Screening for automatic function; (5) Functional analysis (FA); and (6) FBT intervention phase. If steps 1 - 5 determine a participant's challenging behavior serves a social function, Functional Communication Training (FCT) will be administered. If steps 1 - 5 determine a participant's challenging behavior serves an automatic function Competing Stimulus Treatment (CST) will be administered.
  Arms: Functional Behavioral Training
Other: Positive Parenting Strategies-Treatment as Usual — Using the Planned Adaptation approach, to identify proactive adaptations seeking to improve the fit of FBTsIDD with the unique needs of the syndromic IDD population. Triangulating mixed methods data from systematic video observations, questionnaires, and qualitative interviews, then the Framework for Reporting Adaptations and Modifications-Expanded24 (FRAME) will be used to develop a rich understanding of these and any additional adaptations made to the intervention when delivered by non-specialist providers within medical hubs serving syndromic IDD populations.
  Arms: Positive Parenting Strategies-Treatment As Usual

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an adapted, telehealth functional behavioral therapy (FBTsIDD) specifically focused on promoting appropriate communication and behavioral strategies in individuals with syndromic intellectual and developmental disorders.

Participants will be asked to complete virtual study assessments at intake and then on a monthly basis for the duration of 3-6 months. In addition, participants will attend weekly or biweekly virtual intervention visits with a study therapist.

ELIGIBILITY:
Inclusion Criteria:

* Age(s) 2-12 years old at time of enrollment
* Existing genetic syndrome based on clinical or genetic diagnosis and confirmed by medical records
* Documented diagnosis of global developmental delay (GDD) or intellectual disability (ID)
* estimated ID in all ranges
* Disruptive behavior challenges determined to be clinically appropriate for remote, parent-implemented coaching based on clinician determination of acuity of problem behaviors
* Caregiver who is able to consent in English.
* Parent/caregiver available for weekly intervention sessions
* Stable psychosocial and psychiatric treatments 3 months prior to baseline visit.

Exclusion Criteria:

* High levels of aggression that mitigate remote or outpatient treatment as defined by clinician judgement and/or ABC Irritability scores above 20 (i.e., higher level of care needed than provided by study procedures)
* Medical or psychiatric instability that may limit study participation
* Meaningful change in medication or psychosocial interventions 3 months prior to baseline visit
* Limitations in technology access that may hinder participation in remote trial (e.g., declining support provided by study participation)

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression | TO (Baseline), T2 (Month 2), T4 (Month 4), T6 (Month 6)
  Overall functioning will be measured using the Clinical Global Impression for Severity (CGI-S) and Improvement (CGl-I). GCI-S will be recorded at Baseline with CGI-S and CGI-I collected at all determined visits. The CGI provides a rating of the child's global functioning, taking into account all available information (e.g., child's symptoms, behavior, functioning). The CGI-S and CGl-I will be completed by a blinded independent evaluator.

SECONDARY OUTCOMES:
Parent Target Problems (PTP) Inventory | TO (Baseline), T2 (Month 2), T4 (Month 4), T6 (Month 6)
  The Parent Target Problems is a blinded rating provided by an independent evaluator and based on a caregiver interview (30-minutes at baseline; 10- to 15-minutes at follow-visits throughout the study). The independent evaluator will use the PTP interview to record the caregivers' estimate of the frequency of problematic behaviors. From this description, the independent evaluator (blind to treatment assignment) will generate a brief narrative describing the child's problem behaviors and their impact on daily functioning. The evaluator will read this back to the caregiver to provide corrections and/or add any pertinent missing information. This process will continue until the narrative represents an accurate description per caregiver report. Change on the chief concerns determined from interviews are then rated on a 9-point scale (1=normalized, 5=unchanged, 9=disastrous). The PTP has been used to measure outcomes in behavioral intervention trials.
Aberrant Behavior Checklist, Second Edition (ABC-2) | TO (Baseline), T2 (Month 2), T4 (Month 4), T6 (Month 6)
  The Aberrant Behavior Checklist, Second Edition (ABC-2) is a widely-used symptom checklist (completed by caregivers) that measures problematic behavior across five domain subscales: irritability, social withdrawal, stereotypic behavior, hyperactivity/noncompliance, inappropriate speech. Changes in raw scores across each subscale will be tracked against caregiver reports described in the PTP.
Adverse Event Monitoring | TO (Baseline), T1 (Month 1), T2 (Month 2), T3 (Month 3), T4 (Month 4), T5 (Month 5), T6 (Month 6)
  Adverse events will be measured at each time point, and the log used in this study will be based on adverse event logs that have already been developed for other ongoing NIH trials in our center. The adverse event log will include data on any adverse events, the onset date, intensity of event(s), relationship to study (i.e., unrelated through definitely related), end date, outcome, regulatory action taken (if necessary), and whether treatment was required.

CONTACTS AND LOCATIONS:
Locations (1):
- Autism Assessment Research Treatment and Services (AARTS) Center at Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No